CLINICAL TRIAL: NCT03138993
Title: Improving Older Adults' Decision Making for Obstructive Sleep Apnea Treatment (Phase 3)
Brief Title: Improving Older Adults' Decision Making for OSAT
Acronym: eDecide2Rest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Constance Fung, MD, MSHS, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16001482
Record Dates: First submitted 2017-02-14; First posted 2017-05-03 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient decision aid (Active Comparator)
  Interventions: Behavioral: Patient decision aid
- General sleep education (Sham Comparator)
  Interventions: Behavioral: General sleep education

INTERVENTIONS:
Behavioral: Patient decision aid — Web-based patient decision aid plus a paper workbook.
  Arms: Patient decision aid
Behavioral: General sleep education — Web-based information about sleep plus a paper workbook
  Arms: General sleep education

SUMMARY:
This study evaluates the feasibility of conducting a randomized controlled trial that tests a patient decision aid for obstructive sleep apnea in older adults with newly-diagnosed obstructive sleep apnea treated in an outpatient sleep clinic. Half of the participants will use a patient decision aid, while the other half will receive general information about sleep.

DETAILED DESCRIPTION:
Patient decision aids are one strategy for helping older adults make informed decisions about treatments. Patient decision aids improve patients' knowledge about therapies and encourage them to actively weigh the risks and benefits of each therapy.

ELIGIBILITY:
Inclusion Criteria:

1. age >= 60 years
2. diagnosed with obstructive sleep apnea on a sleep study
3. able to read English-language newspaper text (if needed, using contact lens/glasses)
4. able to write words in a paper booklet
5. scheduled for a sleep clinic appointment with a UCLA sleep provider
6. able to attend a sleep educational session prior to sleep clinic appointment

Exclusion Criteria:

1. unable to provide informed consent
2. dementia
3. mild cognitive impairment diagnosis or Mini-Cog score < 3
4. treated for obstructive sleep apnea for > 30 days prior to scheduled sleep education intervention
5. severe physical or mental illness (e.g., hospitalized within past 7 days prior to scheduled sleep education intervention, substance abuse within 90 days of sleep education intervention)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rates | Through study completion, an average of 1 year
  The investigators will measure recruitment rates for our recruitment strategies
Enrollment rates | Through study completion, an average of 1 year
  The investigators will measure enrollment rates

SECONDARY OUTCOMES:
The length of time for completing the intervention session | Through study completion, an average of 1 year
  The investigators will measure the length of time for completing the intervention session

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fung CH, Martin JL, Liang LJ, Hays RD, Col N, Patterson ES, Josephson K, Mitchell MN, Sanchez MC, Aysola R, Song Y, Dzierzewski JM, Huang D, Zeidler M, Alessi C. Efficacy of a patient decision aid for improving person-centered decision-making by older adults with obstructive sleep apnea. J Clin Sleep Med. 2021 Feb 1;17(2):121-128. doi: 10.5664/jcsm.8798. PMID 32955013